CLINICAL TRIAL: NCT00536939
Title: A Randomized, Double-Blind, Phase 2 Trial of Paclitaxel Plus Bevacizumab and Enzastaurin Versus Paclitaxel Plus Bevacizumab and Placebo for Locally Recurrent or Metastatic Breast Cancer
Brief Title: Trial of Paclitaxel, Bevacizumab, and Enzastaurin Versus Paclitaxel, Bevacizumab and Placebo for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been terminated due to slow enrollment
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11396; H6Q-MC-S038 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — enzastaurin; Bevacizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzastaurin + Bevacizumab + Paclitaxel (Experimental): Participants randomized to this arm (Arm A) will receive enzastaurin, paclitaxel and bevacizumab until disease progression.
  Prior to randomization, a safety lead-in will be conducted in 6 participants who will be treated according to Arm A for 2 cycles (1 cycle = 28 days). Only after an acceptable safety analysis of the safety lead-in, will other participants be randomized to Phase 2 (either Arm A or Arm B). In Phase 2, participants from the safety lead-in will continue treatment according to Enzastaurin + Bevacizumab + Paclitaxel (Arm A).
  Interventions: Drug: Enzastaurin; Drug: Bevacizumab; Drug: Paclitaxel
- Bevacizumab + Paclitaxel + Placebo (Placebo Comparator): Participants randomized to this arm (Arm B) will receive bevacizumab, paclitaxel and placebo until disease progression.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Enzastaurin — 1125 milligrams (mg) loading dose on Day 1 of Cycle 1 only then 500 mg oral once daily, until disease progression
  Other Names: LY317615
  Arms: Enzastaurin + Bevacizumab + Paclitaxel
Drug: Bevacizumab — 10 milligrams per kilogram (mg/kg) intravenously, Days 1 and 15 every 28 days, until disease progression
Drug: Paclitaxel — 90 milligrams per square meter (mg/m^2), intravenously, Days 1 ,8, and 15 every 28 days until disease progression
Drug: Placebo — Oral, daily, until disease progression
  Arms: Bevacizumab + Paclitaxel + Placebo

SUMMARY:
The purpose of this study is to determine efficacy and safety of paclitaxel, bevacizumab and enzastaurin versus paclitaxel, bevacizumab, and placebo in participants who are diagnosed with locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have signed an inform consent document
* Have histologic or cytologic diagnosis of breast cancer with evidence of unresectable locally recurrent or metastatic disease
* Have not received any prior chemotherapy for locally recurrent or metastatic disease
* Have not had adjuvant or neoadjuvant taxane therapy within 12 months prior to assignment to study treatment
* Age 18 years or older at time of informed consent

Exclusion Criteria:

* Have any clinical evidence of central nervous system (CNS) metastases
* Have a history of seizure
* Have had a major surgical procedure within 4 weeks prior to assignment to study treatment
* Have had a minor surgical procedure, placement of an access device, or fine needle aspiration within 7 days prior to assignment to study treatment
* Have symptomatic peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galesburg, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goshen, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a safety lead-in prior to randomization. The study was terminated prior to completion of safety lead-in period.
Groups:
- Enzastaurin + Bevacizumab + Paclitaxel: Safety Lead-in Period: Enzastaurin 1125 milligrams (mg) loading dose (total nine 125-mg tablets: 3 tablets, 3 times daily) administered orally, only on Day 1 of Cycle 1, followed by 500 mg (four 125-mg tablets) administered orally, once daily in a 28-day cycle plus bevacizumab 10 milligrams per kilogram (mg/kg) administered intravenously on Days 1 and 15 of every 28-day cycle plus paclitaxel 90 milligrams per square meter (mg/m^2) administered intravenously on Days 1, 8 and 15 of every 28-day cycle. Participants were to receive enzastaurin, bevacizumab and paclitaxel for 2 cycles (1 cycle = 28 days).
  Randomization Period: Participants were to receive the same treatment as administered during the safety lead-in period. Treatment was to continue until there was evidence of disease progression or intolerable toxicity.
- Bevacizumab + Paclitaxel + Placebo: Safety lead-in Period: No treatment
  Randomization Period: Participants were to receive bevacizumab 10 mg/kg administered intravenously on Days 1 and 15 of every 28-day cycle plus paclitaxel 90 mg/m^2 administered intravenously on Days 1, 8 and 15 of every 28-day cycle plus placebo loading dose administered orally (total 9 tablets: 3 tablets, 3 times daily) only on Day 1 of Cycle 1, followed by oral administration once daily in a 28-day cycle. Treatment was to continue until there was disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | Enzastaurin + Bevacizumab + Paclitaxel | Bevacizumab + Paclitaxel + Placebo
Started | 2 | 0
Entered Safety lead-in | 2 | 0
Randomized | 0 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Complicating Disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Enzastaurin + Bevacizumab + Paclitaxel
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of study enrollment to the first date of objectively determined progressive disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST version 1.0). PD is ≥20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. For participants not known to have died and who did not have PD, PFS was censored at the date of the last progression-free assessment. For participants who received subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to disease progression or death, PFS was censored at the date of last progression-free assessment prior to the initiation of post-discontinuation systemic anticancer therapy. No participant completed a full cycle of therapy and thus no formal analysis was performed.
Time Frame: Baseline to measured PD (up to 15 days)
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Enzastaurin + Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR), assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST version 1.0). CR was defined as the disappearance of all tumor lesions; PR was defined as either ≥30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions. In either case of PR, no new lesions should have appeared. The percentage of participants with ORR was calculated as a total number of participants with CR or PR from the start of study treatment until disease progression or recurrence divided by the total number of participants treated, then multiplied by 100. No participant completed a full cycle of therapy and thus no formal analysis was performed.
Time Frame: Baseline to measured Progressive disease (up to 15 days)
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Enzastaurin + Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Any Serious AEs (SAEs)
Description: A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline to study completion (Day 15) plus 30-day safety follow-up
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- Enzastaurin + Paclitaxel + Bevacizumab: Safety Lead-in Period: Enzastaurin 1125 milligrams (mg) loading dose (total nine 125-mg tablets: 3 tablets, 3 times daily) administered orally, only on Day 1 of Cycle 1, followed by 500 mg (four 125-mg tablets) administered orally, once daily in a 28-day cycle plus bevacizumab 10 milligrams per kilogram (mg/kg) administered intravenously on Days 1 and 15 of every 28-day cycle plus paclitaxel 90 milligrams per square meter (mg/m^2) administered intravenously on Days 1, 8 and 15 of every 28-day cycle. Participants were to receive enzastaurin, bevacizumab and paclitaxel for 2 cycles (1 cycle = 28 days).
  Randomization Period: Participants were to receive the same treatment as administered during the safety lead-in period. Treatment was to continue until there was evidence of disease progression or intolerable toxicity.
Arm/Group | Enzastaurin + Paclitaxel + Bevacizumab
Number analyzed (Participants) | 2
Participants
  Adverse Events (AEs) | 2
  Serious Adverse Events (SAEs) | 0

ADVERSE EVENTS:
Arm/Group | Enzastaurin + Bevacizumab + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin + Bevacizumab + Paclitaxel (N=2)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow enrollment and competing studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days